CLINICAL TRIAL: NCT00922584
Title: A Phase II Study of Sorafenib (BAY 43-9006®) in Patients With Relapsed Advanced Non-Small Cell Lung Cancer(NSCLC) After Failure of Epidermal Growth Factor Receptor-tyrosine Kinase Inhibitor (EGFR-TKI)Treatment
Brief Title: Sorafenib Treatment in Non-Small Cell Lung Cancer After Failure of Epidermal Growth Factor Receptor-tyrosine Kinase Inhibitor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese Society of Lung Cancer (Other)
Responsible Party: Principal Investigator, Yi-Long Wu, Director of Chinese Society of Lung Cancer/Chief of Lung Cancer Research Institute & Cancer Center/Vice President of Guangdong General hospital, Chinese Society of Lung Cancer
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-TONG0805
Record Dates: First submitted 2009-06-09; First posted 2009-06-17 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: non-small cell lung cancer; Sorafenib; targeted therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sorafenib (Experimental): Patients with stage IIIB/IV NSCLC who failed EGFR-TKI therapy will receive oral sorafenib 400 mg twice daily until disease progression or unacceptable toxicity.
  Interventions: Drug: sorafenib (Nexavar)

INTERVENTIONS:
Drug: sorafenib (Nexavar) — oral sorafenib 400 mg, twice daily, until disease progression or unacceptable toxicity

SUMMARY:
This trial's aim is to evaluate the efficacy and toxicity of sorafenib in relapsed advanced Non-Small Cell Lung Cancer (NSCLC) after failure of epidermal growth factor receptors-tyrosine kinase inhibitor (EGFR-TKI) treatment and to explore the correlation between clinical outcomes and biochemical modulation of signal transduction pathways.

DETAILED DESCRIPTION:
Sorafenib, an oral multi-kinase inhibitor, targets the Raf/MEK/ERK pathway at the level of Raf kinase and VEGF receptor tyrosine kinases, and has shown efficacy against NSCLC in Phase I/II trials. Because the targets of sorafenib are different from that of EGFR-TKI, it is reasonable for sorafenib to treat relapsed advanced NSCLC after failure of EGFR-TKI treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological documented stage IIIB (not amenable for radical regional therapy) or stage IV NSCLC. The pathological diagnosis must be adenocarcinoma with or without bronchioalveolar carcinoma. Sputum cytology alone is excluded.
* Recurrent or progressive disease after prior one EGFR-TKI treatment. The patient must have stopped the EGFR-TKI treatment for at least two weeks. The response to EGFR-TKI should be partial response or complete response or stable disease (the duration of stable disease should be more than 3 months). Patients who had never received chemotherapy or received one regimen chemotherapy before EGFR-TKI are eligible.
* Prior surgery, including palliative surgery, is permitted if performed 4 weeks before the start of study treatment and the patient is fully recovered.
* Prior localized radiotherapy 4 weeks before the start of study is permitted if it was not administered to target lesions selected for this study, unless progression of the selected target lesions within the radiation portal is documented. Patient has recovered from CTCAE grade 3/4 toxicity of radiotherapy. Palliative radiotherapy within 4 weeks of start of study is also permitted.
* Age > 18 years.
* ECOG Performance Status of 0, 1,or 2. Life expectancy of at least 3 months. Measurable disease, according to the RECIST, the presence of at least one uni-dimensional measurable lesion with longest diameter > 20 mm by conventional techniques or > 10 mm by spiral CT scan.
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:
* Hemoglobin > 9.0 g/dl
* Platelet count > 75x109/L
* Total bilirubin ≤ 1.5 x upper limit of normal
* ALT and AST < 2.5 x upper limit of normal without liver metastasis, ALT and AST < 5 x upper limit of normal with liver metastasis.
* International normalized ratio (INR) ≤ 1.5 x the upper limit of normal and prothrombin time (PT) ≤ 1.5 x the upper limit of normal. Patients who are being therapeutically anticoagulated with an agent such as Coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists.
* Serum creatinine < 1.5 x upper limit of normal.

Exclusion Criteria:

* Patients who are currently enrolled in, are eligible for, or have access to, any other sorafenib clinical trial.
* Mixed small cell and non-small cell lung cancer histology. Other pathological types of NSCLC than adenocarcinoma and bronchioloalveolar cell carcinoma.
* Failure of EGFR-TKI is due to toxicity.
* Prior with exposure to biotherapy, immunotherapy within 4 weeks of study entry.
* Prior exposure to sorafenib or other agents targeting the Ras/MARK pathway or VEGFR.
* Any unresolved toxicity more than CTCAE grade 2 from previous anti-cancer therapy.
* Patients with cardiac arrhythmias greater than grade 1 NCI CTCAE, Version 3.0(Conduction abnormality and supraventricular arrhythmia present but patient is asymptomatic; intervention not indicated, palpitations present and QTC > 0.45-0.47 second); however, patients with grade 2 atrial fibrillation may be included.
* Significant cardiovascular event: congestive heart failure > NYHA class 2; unstable angina, active CAD (myocardial infarction more than 6 months prior to study entry is allowed); serious cardiac arrhythmia requiring anti-arrythmic therapy (beta blockers or digoxin are permitted) or uncontrolled hypertension.
* Any disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of any study medication (sorafenib) or that might affect the interpretation of the results or render the subject at high risk from treatment.
* Central nervous system (CNS) tumor or metastatic tumor.
* Clinically significant gastrointestinal bleeding within 30 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2008-12; Primary Completion 2012-01 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Disease control rate (CR+PR+SD) | 1 year

SECONDARY OUTCOMES:
Response duration | 2 years
time-to-progression | 2 years
progression free survival | 2 years
overall survival | 2 years
safety profile | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Wu Yi Long, Professor, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- WuYiLong, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhou Q, Zhou CC, Chen GY, Cheng Y, Huang C, Zhang L, Xu CR, Li AW, Yan HH, Su J, Zhang XC, Yang JJ, Wu YL. A multicenter phase II study of sorafenib monotherapy in clinically selected patients with advanced lung adenocarcinoma after failure of EGFR-TKI therapy (Chinese Thoracic Oncology Group, CTONG 0805). Lung Cancer. 2014 Mar;83(3):369-73. doi: 10.1016/j.lungcan.2013.12.014. Epub 2014 Jan 5. PMID 24440279